CLINICAL TRIAL: NCT06575998
Title: The Treatment of Insomnia in Primary Care: Evaluating and Improving Compliance to Clinical Practice Guidelines
Brief Title: Insomnia in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, menumans, Prof. dr. M.E. Numans, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N24.054; 80-83910-98-1158 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2024-08-16; First posted 2024-08-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Insomnia
Keywords: Primary Care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The cluster randomization trial involves two randomization procedures. Firstly, on primary care practice level, practices will be randomized to intervention practice or control practice. Secondly, patients in the intervention practices will be randomized to pro-active identification or no identification. Pro-actively identified insomnia patients will be reported back to the PCP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training with pro-active identification (Experimental): For detailed description of the intervention, see the separate section on interventions.
  Interventions: Other: Training; Other: Pro-active identification
- Training without pro-active identification (Experimental): For detailed description of the intervention, see the separate section on interventions.
  Interventions: Other: Training
- Control (No Intervention): Care as usual according to national applicable primary guide guidelines.

INTERVENTIONS:
Other: Training — A 4-hour training for PCPs consisting of an onsite training, an e-learning and a webinar on the treatment of insomnia.
  Arms: Training with pro-active identification; Training without pro-active identification
Other: Pro-active identification — Pro-active identification of patients with clinical insomnia symptoms. Patients receiving care from the participating practices will be asked to fill-out the Insomnia Severity Index (ISI).The ISI is used to identify patients with clinical insomnia symptoms in the general practice. Trained practices will receive feedback on the ISI for half of the patients with clinical symptoms according to the ISI.
  Arms: Training with pro-active identification

SUMMARY:
The goal of this clinical trial is to learn if training primary care providers on treatment of insomnia can improve insomnia symptoms in patients. Researchers will compare insomnia symptoms of patients receiving care from trained practices with patients receiving care from control practices (providing care-as-usual), to see if the training helps to provide improved insomnia care. Participants will be asked to complete four questionnaires and some participants will be invited for an insomnia consultation in primary care by their primary care providers (PCP).

ELIGIBILITY:
Inclusion criteria for a patient to be eligible to participate in this study:

1. Patient registered with a participating primary care facility and willing to provide informed consent AND
2. Survey confirmed presence of insomnia symptoms at least 3 times a week during at least the last 3 weeks AND
3. Survey shown increased score on the Insomnia Severity Index (ISI ≥ 11) AND
4. Survey shown interference with daily functioning on the Insomnia Severity Scale.

Exclusion criteria:

Patients meeting any of the following criteria in the survey will be excluded from participation in this study:

1. Shift work for individuals awakening outside the hours 4:00 A.M. and 10:00 A.M. or going to bed outside the hours of 8:00 P.M. and 2:00 A.M. more than twice a week
2. Other sleep-wake disorders including chronic obstructive sleep apnea, bruxism and narcolepsy, restless leg syndrome and parasomnia.
3. Current pregnancy
4. Presence of epilepsy, schizophrenia, bipolar disorder, post-traumatic stress disorder or dementia in medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported insomnia symptoms using the Insomnia Severity Index (ISI) | From baseline to measurements at 2, 6 and 12 months
  Change is measured linearly using the Insomnia Severity Index. Scores range from 0 to 28 points in which higher scores represent a worse outcome. Secondly, the categorically defined treatment response is established 2 months after baseline questionnaire (remission = ISI score < 11, ISI score reduction ≥ 8).

SECONDARY OUTCOMES:
Patient reported non-pharmacological 'sleep consultation' | 12 months after baseline questionnaire
  Patient report of a sleep consultation (survey answer yes/no) combined with patient reported sleep medication use (survey answer yes/no).
Report by the PCP of a non-pharmacological 'sleep consultation' | 12 months after baseline questionnaire
  PCP reported sleep consultation (survey answer yes/no) combined with PCP reported sleep medication use (survey answer yes/no).
Change in patient reported depression symptoms | From baseline to measurements at 2, 6 and 12 months
  Measured linearly using the Patient Health Questionnaire-9 (PHQ-9). Scores range from 0 to 27 points in which higher scores represent a worse outcome.
Change in patient reported anxiety symptoms | From baseline to measurements at 2, 6 and 12 months
  Measured linearly using the General Anxiety Disorder Questionniare (GAD-7). Scores range from 0 to 21 points in which higher scores represent a worse outcome.
Change in patient reported general health status | From baseline to measurements at 2, 6 and 12 months
  Measured with the Short Form-36 questionnaire (SF-36). Scores represent the percentage of total possible score achieved, ranging from 0 to 100. A higher score represents a better outcome.
Change in report of sleep medication use | From baseline to measurements at 2, 6 and 12 months
  Patient reported use of sleep medication in the past two weeks (survey answer yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis O. Mook-Kanamori, Principal Investigator — Leiden University Medical Center (LUMC); Rutger A. Middenburg, Principal Investigator — Leiden University Medical Center (LUMC); Mattijs E. Numans, Principal Investigator — Leiden University Medical Center (LUMC)
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Due to the nature of the study blinding is not possible. Therefore, the data contains privacy sensitive information and only restricted access may be granted for unidentifiable parts of the data. It has yet to be decided which data can be acquired through restricted access.